CLINICAL TRIAL: NCT04853914
Title: Evaluation of the Safety of the Treatment of Benign Prostatic Hyperplasia by High Intensity Focused Ultrasound.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/F/20.09
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Adenoma; Prostate; HIFU; Mini-invasive treatment
MeSH Terms: conditions — Prostatic Hyperplasia; Adenoma

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, mono-centric, non-controlled, non-randomized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIFU intervention (Experimental): Patients will benefit of an HIFU treatment of their Benign Prostatic Hyperplasia.
  Interventions: Device: HIFU treatment

INTERVENTIONS:
Device: HIFU treatment — HIFU treatment of Benign Prostatic Hyperplasia

SUMMARY:
Prostate adenoma or benign prostatic hypertrophy (BPH) is a benign disease of the prostate gland. It results in an increase in the volume of the prostate area located in contact with the urethra. Compression of the prostatic urethra by the adenoma can cause lower urinary tract disorders.

The classic treatments in case of failure of medical treatment are endoscopic resection of the prostate and adenomectomy, but these techniques are characterized by a significant hemorrhagic risk that may require transfusions and prolonged hospitalization.

Minimally invasive treatments with low morbidity have been developed to overcome these drawbacks. They allow to propose a therapeutic solution adapted to patients: not tolerating their medical treatment, wishing to keep antegrade ejaculation, elderly and/or frail, at risk of bleeding, wishing an ambulatory treatment, refusing the conventional surgical techniques.

The Focal One® device was developed to treat prostate cancer using ultrasound energy. This energy is delivered through a probe placed in your rectum. Connected to this probe, an ultrasound machine will allow your doctor to see precisely which part of your prostate is being treated. By heating the prostate tissue to a very high temperature in one treatment session, the energy delivered will then destroy the tissue. Ultrasound guidance coupled with the localized nature of the treatment allows the targeted area to be treated while respecting the prostate tissue and structures adjacent to the prostate and thus reducing side effects.

Treatment of prostate adenoma with HIFU would allow for localized destruction to reduce prostate volume. The reduction of the compression of the prostatic urethra thus obtained would allow an improvement of the urinary disorders. The treatment is performed transrectally under real-time ultrasound control, which allows the adjacent structures to be respected, thus preserving antegrade ejaculation and limiting the side effects.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years of age,
* BPH greater than 30 cc confirmed by endorectal ultrasound
* IPSS score > 7, Qol-IPSS > 2, IIEF-5 score > 11
* Qmax < 15 ml/s or urinary retention (in indwelling catheter, self-catheterization, or with an RPM > 300 cc).
* In failure or intolerance of drug treatment(s) for BPH
* negative cytobacteriological examination of the urine

Exclusion Criteria:

* Prostate volume > 80 ml
* Presence of a median lobe
* Men allergic to latex
* Contraindication to the insertion of a transrectal HIFU probe: rectal fistula, anal or rectal fibrosis, or other abnormalities
* History of prostate surgery
* History of prostate radiation therapy
* History of bladder cancer
* Current anti-coagulant treatment with a stopping window that cannot exceed 48 hours at the time of the HIFU procedure
* Presence of a urinary tract fistula
* History of inflammatory bowel disease
* Ongoing urogenital infection
* Neurological bladder pathology
* History of urethral stenosis
* Confirmed or suspected prostate cancer
* Contraindication to surgery (including anesthesia)
* Contraindication to pelvic MRI
* Presence of metallic implants or stents in the urethra
* Presence of prostatic calcification whose location interferes with HIFU treatment
* Patients with renal failure with a GFR <35ml/min

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The safety of HIFU treatment will be assessed by analyzing adverse events (serious and non-serious) reported during follow-up. | 3 months

SECONDARY OUTCOMES:
Evaluation of treatment performance by maximum urine output (Qmax) | 1 and 3 months
Evaluation of treatment performance by residual post-void volume (RPM) | 1 and 3 months
Evaluation of voiding symptomatology with IPSS questionnaire | 1 and 3 months
Evaluation of quality of urinary life with Qol-IPSS score | 1 and 3 months
Evaluation of quality of erection with IIEF-5 questionnaire | 1 and 3 months
Evaluation of ejaculation quality with MSHQ-SF questionnaire | 1 and 3 months
Evaluation of continence with ICIQ-SF questionnaire | 1 and 3 months
Evaluation of the global impression of improvement scale with PGI-1 questionnaire | 1 and 3 months
Evaluation of the change in the PSA rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Codas-Duarte, DR, Principal Investigator — HCL
Locations (1):
- Hopital Edouard Herriot, service d'urologie, Lyon, France

IPD SHARING:
Plan to Share IPD: No